CLINICAL TRIAL: NCT04357158
Title: Breath analysiS as an Additional Test for ColoREctal cancEr screeNing to rEduce the Number of unnecessaRy Colonoscopies
Acronym: SCREENER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: '2020-6184'
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer; Polyp of Colon; Colorectal Neoplasms
Keywords: Volatile organic compounds; VOC; Colorectal cancer; Advanced adenoma; Breath test; Electronic nose; eNose; Aeonose
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Intervention Model Description: This is a multicenter prospective cohort study in participants eligible for colonoscopy with suspicion for (pre)malignant lesions of the colon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients referred for colonoscopy (Other)
  Interventions: Device: AeonoseTM

INTERVENTIONS:
Device: AeonoseTM — All participants will be asked to breathe into an electronic nose (eNose, the AeonoseTM, The eNose Company, Zutphen, the Netherlands) for 5 minutes during the pre-colonoscopy intake and just prior to the procedure to assess reproducibility (with >2 weeks in between).

SUMMARY:
In the past decade, the demand for colonoscopy procedures has increased significantly since the introduction of population-based colorectal cancer (CRC) screening in many western countries. Post-polypectomy surveillance will increase the number of colonoscopy procedures conducted each year even further. The invasive nature of colonoscopy and the associated health-care costs warrant the development of a new non-invasive test to reduce the number of unnecessary colonoscopies.

These days, many countries use a non-invasive fecal test for CRC screening which is easy to perform at home, but test characteristics such as sensitivity and specificity are suboptimal. Multiple studies have already shown that volatile organic compound (VOC) analysis has a high diagnostic accuracy for CRC and Advanced Adenomas. An additional VOC analysis, for example through breath testing, in patients with a positive fecal immunochemical test (FIT) may reduce the number of unnecessary colonoscopies.

The aim of this study is to validate the diagnostic accuracy of the AeonoseTM to distinguish patients with CRC from healthy controls, and to assess reproducibility of test results.

DETAILED DESCRIPTION:
Rationale: An electronic nose (eNose) is an artificial olfactory system that analyses volate organic compounds (VOCs) in exhaled breath. Exhaled human breath is mainly composed of inorganic compounds, inert gases and VOCs. VOCs are exhaled in very low concentrations and reflect pathological processes such as inflammation, oxidation, infection and neoplasms. The perspective is that metabolic and biochemical processes in several pathological situations cause different endogenous VOCs to arise, were they can serve as non-invasive biomarkers for certain diseases.

Primary objective: To evaluate if the use of an additional breath test (AeonoseTM) for patients with a positive FIT-test can reduce the number of unnecessary colonoscopies.

Secondary objectives:

1. External validation of results for CRC and (advanced) adenoma detection established in a previous studies (second study not yet published). (15)
2. To evaluate if VOC profiles in breath are similar at two different time points.
3. Acceptance rate of using the AeonoseTM device for VOC analysis in participating patients.

Study population: Patients between the ages of 55 and 75 years old with a positive FIT-test referred for a colonoscopy procedure.

Estimated sample size: 750 participants

Intervention: Participants will be asked to breath through the AeonoseTM for 5 minutes during pre-colonoscopy intake and just prior to the procedure to assess reproducibility (with >2 weeks in between). There are no risks, nor benefits for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 55 and 75 years referred for a colonoscopy procedure after a positive FIT test, according to the population based CRC screening program in the Netherlands

Exclusion Criteria:

* Prior surgical resection of any portion of the colon
* History of any type of malignancy, not including squamous cell carcinoma (SCC) and basal cell carcinoma (BCC)
* Current active colitis or history of polyposis syndrome

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy in distinguishing colorectal carcinoma from healthy controls | 12 months
  The diagnostic accuracy, in terms of sensitivity and specificity, of the AeonoseTM in distinguishing between patients with and without CRC.

SECONDARY OUTCOMES:
Diagnostic accuracy in distinguishing advanced adenoma from healthy controls | 12 months
  Sensitivity and specificity
Reproducibility | 12 months
  The variation in VOC analysis results between two separate time points. The binary results from the eNose analysis will be presented in a scatterplot and a receiver operating characteristics curve (ROC-curve). Cohen's kappa statistic will be applied to determine interobserver agreement between the eNose results of 2 different timepoints (>2 weeks apart)
Acceptance rate | 12 months
  The acceptance rate of using the AeonoseTM in participating patients.

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Siersema, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van Riswijk MLM, van Keulen KE, Tan ACITL, Schrauwen RWM, de Vos Tot Nederveen Cappel WH, Siersema PD; eNose CRC study group. Research Communication: Breath Testing for Colorectal Cancer Detection in Patients With a Positive Fecal Immunochemical Test: A Multicentre Prospective Cross-Sectional Study With External Validation. Aliment Pharmacol Ther. 2025 Jul;62(2):208-213. doi: 10.1111/apt.70207. Epub 2025 Jun 3. PMID 40459533
- [Derived] van Riswijk MLM, van Tintelen BFM, Lucas RH, van der Palen J, Siersema PD. Overcoming methodological barriers in electronic nose clinical studies, a simulation data-based approach. J Breath Res. 2025 May 9;19(3). doi: 10.1088/1752-7163/add291. PMID 40306296